CLINICAL TRIAL: NCT01444287
Title: Daytime Corneal Swelling During Wear of Narafilcon B Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-0918 (JKN 0927)
Record Dates: First submitted 2011-09-27; First posted 2011-09-30 (Estimated); Results first posted 2014-05-30 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2015-05

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Spectacles No Lenses (Placebo Comparator): Assigned in random order during one of four 8 hour sessions on four separate days, in one of 24 possible order combinations.
  Interventions: Other: Spectacles
- narafilcon B (Experimental): Assigned in random order during one of four 8 hour sessions on four separate days, in one of 24 possible order combinations.
  Interventions: Device: narafilcon B
- polymacon (Active Comparator): Assigned in random order during one of four 8 hour sessions on four separate days, in one of 24 possible order combinations.
  Interventions: Device: Polymacon
- lotrafilcon A (Active Comparator): Assigned in random order during one of four 8 hour sessions on four separate days, in one of 24 possible order combinations.
  Interventions: Device: Lotrafilcon A

INTERVENTIONS:
Device: narafilcon B — test product
  Arms: narafilcon B
Device: Polymacon — marketed product
  Arms: polymacon
Device: Lotrafilcon A — marketed product
  Arms: lotrafilcon A
Other: Spectacles — None - subject used own spectacles
  Arms: Spectacles No Lenses

SUMMARY:
The purpose of this research is to measure daytime open-eye response to wearing of narafilcon B lenses.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age (i.e. ≥ 18 years).
* Be mentally competent, willing and able to sign a written informed consent form.
* Have contact lens distance sphere requirement in the range -1.00D to -6.00D.
* Have spectacle astigmatism <1.25D in each eye.
* Currently wear soft contact lenses (for at least 6 months prior to the trial) with documentation of current prescription.
* Have normal eyes with no evidence of abnormality or disease. For the purpose of this study a normal eye is defined as one having: i) no evidence of lid abnormality or infection; ii) no conjunctival abnormality or infection; iii) no clinically significant slit lamp findings (i.e, edema, staining, scarring, vascularization, infiltrates or abnormal opacities); iv) no other active ocular disease.

Exclusion Criteria:

* Required concurrent ocular medication.
* Any systemic illness which would contra-indicate lens wear or the medical treatment of which would affect vision or successful lens wear.
* Eye injury or surgery within eight weeks immediately prior to enrollment for this study.
* Abnormal lacrimal secretions.
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Keratoconus or other corneal irregularity.
* Pregnancy, lactating or planning a pregnancy at the time of enrollment.
* Participation in any concurrent clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noel Brennan, McOptom PhD, Principal Investigator — Coles-Brennan Pty Ltd
Locations (1):
- Coles-Brennan Pty Ltd, Hawthorn, Victoria, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 22 subjects enrolled to the study, all completed the four experimental sessions.
Groups:
- All Study Participants: Assigned in random order during one of four 8 hour sessions on four separate days, in one of 24 possible order combinations. The four arms were Spectacles (no contact lenses), Narafilcon B, Polymacon A, and Lotrafilcon A, in random order during the sessions.
Period: Period 1
Arm/Group | All Study Participants
Started | 22
Completed | 22
Not Completed | 0
Period: Period 2
Arm/Group | All Study Participants
Started | 22
Completed | 22
Not Completed | 0
Period: Period 3
Arm/Group | All Study Participants
Started | 22
Completed | 22
Not Completed | 0
Period: Period 4
Arm/Group | All Study Participants
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: Subjects who were enrolled and randomized to a trial arm.
Arm/Group | All Subjects
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 8
Region of Enrollment [Number; unit: participants]
  Australia | 22

OUTCOME MEASURES:

1. Primary Outcome: Corneal Thickness
Description: Percentage of corneal swelling (positive value) or deswelling (negative value) measured with Haag-Streit pachymetry equipment in microns, reported as a percent.
Time Frame: After 8 hours of contact lens wear
Population: Subjects are those enrolled and randomized to a trial arm.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Spectacles No Lenses | Narafilcon B | Polymacon | Lotrafilcon A
Number analyzed (Participants) | 22 | 22 | 22 | 22
Percent Change | -0.35 (0.15) | -0.99 (0.18) | 0.75 (0.21) | -1.02 (0.23)
Statistical Analysis 1: Comparison: Spectacles No Lenses vs Narafilcon B; Ho: No Lenses (control) - narafilcon B (test) = 0. Ha: No Lenses (control) - narafilcon B (test) ≠ 0; Test type: Superiority or Other; p = 0.0035, Mixed Models Analysis; Mean Difference (Final Values) = 0.636, Standard Error of Mean 0.2093 — The mean difference is calculated as: Control-Test
Statistical Analysis 2: Comparison: Narafilcon B vs Polymacon; Ho: Polymacon (+ control) - Narafilcon B (test) = 0. Ha: Polymacon (+ control) - Narafilcon B (test) ≠ 0; Test type: Superiority or Other; p = 0.0000, Mixed Models Analysis; Mean Difference (Final Values) = 1.743, Standard Error of Mean 0.2093 — The mean difference is calculated as: Control - Test
Statistical Analysis 3: Comparison: Narafilcon B vs Lotrafilcon A; Ho: lotrafilcon A (control) - narafilcon B (test) = 0. Ha: lotrafilcon A (control) - narafilcon B (test) ≠ 0; Test type: Superiority or Other; p = 0.8957, Mixed Models Analysis; Mean Difference (Final Values) = -0.0275, Standard Error of Mean 0.2093 — The mean difference is calculated as: Control-Test

2. Primary Outcome: Endothelial Blebs
Description: Corneal images captured with equipment are measured, manually outlined to estimate total bleb area from 0 to 100%. This is measured as a change in percentage after 20 minutes compared to the value prior to lens wear (baseline).
Time Frame: baseline, after 20 minutes of treatment conditions
Measure: Mean (Standard Error); unit: percentage of bleb area
Arm/Group | Spectacles No Lenses | Narafilcon B | Polymacon | Lotrafilcon A
Number analyzed (Participants) | 22 | 22 | 22 | 22
percentage of bleb area | -0.13 (0.31) | 0.49 (0.23) | 0.41 (0.40) | 0.38 (0.41)
Statistical Analysis 1: Comparison: Spectacles No Lenses vs Narafilcon B; Ho: No Lenses (control) - narafilcon B (test) = 0. Ha: No Lenses (control) - narafilcon B (test) ≠ 0; Test type: Superiority or Other; p = 0.0692, Mixed Models Analysis; Mean Difference (Final Values) = -0.0057, Standard Error of Mean 0.0031 — The mean difference is calculated as: Control-Test
Statistical Analysis 2: Comparison: Narafilcon B vs Polymacon; Ho: Polymacon (+ control) - Narafilcon B (test) = 0. Ha: Polymacon (+ control) - Narafilcon B (test) ≠ 0; Test type: Superiority or Other; p = 0.7301, Mixed Models Analysis; Mean Difference (Final Values) = -0.0011, Standard Error of Mean 0.0032 — The mean difference is calculated as: Control-Test
Statistical Analysis 3: Comparison: Narafilcon B vs Lotrafilcon A; Ho: lotrafilcon A (control) - narafilcon B (test) = 0. Ha: lotrafilcon A (control) - narafilcon B (test) ≠ 0; Test type: Superiority or Other; p = 0.8055, Mixed Models Analysis; Mean Difference (Final Values) = -0.0008, Standard Error of Mean 0.0032 — The mean difference is calculated as: Control-Test

3. Primary Outcome: Limbal Redness
Description: Scale of 0 to 4, where 0=none and 4= severe redness. Measure reported as a comparison of 8 hours of wear to baseline with the difference being reported.
Time Frame: Baseline, After 8 hours of treatment conditions
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Spectacles No Lenses (Control); Narafilcon B (Test); Polymacon (+ Control); Lotrafilcon A (Control): Assigned in random order during one of four 8 hour sessions on four separate days, in one of 24 possible order combinations.
Arm/Group | Spectacles No Lenses (Control) | Narafilcon B (Test) | Polymacon (+ Control) | Lotrafilcon A (Control)
Number analyzed (Participants) | 22 | 22 | 22 | 22
units on a scale | -0.03 (0.06) | -0.04 (0.5) | 0.64 (0.10) | 0.13 (0.08)
Statistical Analysis 1: Comparison: Spectacles No Lenses (Control) vs Narafilcon B (Test); Ho: No Lenses (control) - narafilcon B (test) = 0. Ha: No Lenses (control) - narafilcon B (test) ≠ 0; Test type: Superiority or Other; p = 0.9127, Mixed Models Analysis; Mean Difference (Final Values) = 0.0122, Standard Error of Mean 0.1111 — The mean difference is calculated as: Control-Test
Statistical Analysis 2: Comparison: Narafilcon B (Test) vs Polymacon (+ Control); Ho: Polymacon (+ control) - Narafilcon B (test) = 0. Ha: Polymacon (+ control) - Narafilcon B (test) ≠ 0; Test type: Superiority or Other; p = 0.0000, Mixed Models Analysis; Mean Difference (Final Values) = 0.6864, Standard Error of Mean 0.1098 — The mean difference is calculated as: Control-Test
Statistical Analysis 3: Comparison: Narafilcon B (Test) vs Lotrafilcon A (Control); Ho: lotrafilcon A (control) - narafilcon B (test) = 0. Ha: lotrafilcon A (control) - narafilcon B (test) ≠ 0; Test type: Superiority or Other; p = 0.1256, Mixed Models Analysis; Mean Difference (Final Values) = 0.1705, Standard Error of Mean 0.1098 — The mean difference is calculated as: Control-Test

4. Secondary Outcome: Overall Comfort
Description: Patient reported subjective comfort of lenses or spectacles (range 0-100, where 100 is best).
Time Frame: after 8 hours
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Spectacles No Lenses (Control) | Narafilcon B (Test) | Polymacon (+ Control) | Lotrafilcon A (Control)
Number analyzed (Participants) | 22 | 22 | 22 | 22
units on a scale | 96.0 (1.3) | 96.1 (1.0) | 78.3 (5.1) | 80.7 (4.4)
Statistical Analysis 1: Comparison: Spectacles No Lenses (Control) vs Narafilcon B (Test); Ho: No Lenses (control) - narafilcon B (test) = 0. Ha: No Lenses (control) - narafilcon B (test) ≠ 0; Test type: Superiority or Other; p = 0.9892, Mixed Models Analysis; Mean Difference (Final Values) = -0.0688, Standard Error of Mean 5.044 — The mean difference is calculated as: Control-Test
Statistical Analysis 2: Comparison: Narafilcon B (Test) vs Polymacon (+ Control); Ho: Polymacon (+ control) - Narafilcon B (test) = 0. Ha: Polymacon (+ control) - Narafilcon B (test) ≠ 0; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis; Mean Difference (Final Values) = -17.75, Standard Error of Mean 4.984 — The mean difference is calculated as: Control-Test
Statistical Analysis 3: Comparison: Narafilcon B (Test) vs Lotrafilcon A (Control); Ho: lotrafilcon A (control) - narafilcon B (test) = 0. Ha: lotrafilcon A (control) - narafilcon B (test) ≠ 0; Test type: Superiority or Other; p = 0.0030, Mixed Models Analysis; Mean Difference (Final Values) = -15.37, Standard Error of Mean 4.984 — The mean difference is calculated as: Control-Test

ADVERSE EVENTS:
Groups:
- Polymacon A; Lotrafilcon A: Assigned in random order during one of four 8 hour sessions on four separate days, in one of 24 possible order combinations.
Arm/Group | Spectacles No Lenses | Narafilcon B | Polymacon A | Lotrafilcon A
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days